CLINICAL TRIAL: NCT05115292
Title: A First-in-Human, Multicenter, Open-label, Phase 1 Dose-Escalation and Cohort Expansion Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BJ-005 in Patients With Advanced Solid Tumor or Lymphoma
Brief Title: A First-in-Human, Phase 1 Dose-Escalation and Cohort Expansion Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of BJ-005 in Patients With Advanced Solid Tumor or Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BJ Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BJ-005-01-001US
Record Dates: First submitted 2021-10-20; First posted 2021-11-10 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Advanced Solid Tumor or Lymphoma
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm1 (Experimental): BJ-005 dose escalation
  Interventions: Biological: BJ-005
- Arm 2 (Experimental): BJ-005 cohort expansion
  Interventions: Biological: BJ-005

INTERVENTIONS:
Biological: BJ-005 — dosed with intravenous infusion

SUMMARY:
This is a first-in-human, Phase 1 study to evaluate the safety, tolerability, and pharmacokinetics of BJ-005 in patients with advanced solid tumor or lymphoma. BJ-005 is a recombinant bifunctional molecule, composed of a humanized anti-PD-L1 IgG1 monoclonal antibody (mAb) fused with a portion of the extracellular domain of human TGF-β receptor II (TGF-βRII).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years.
2. Willing and able to provide signed and dated informed consent prior to any study-related procedures and willing and able to comply with all study procedures.
3. Histologically or cytologically confirmed advanced solid tumors or lymphoma
4. Measurable or evaluable disease per RECIST v1.1
5. ECOG performance status 0 or 1
6. Life expectancy ≥3 months
7. Adequate hepatic function
8. Calculated creatinine clearance (CrCL) > 50 mL/min (Cockroft-Gault Equation)
9. Adequate Hematological function
10. Prothrombin time, international normalized ratio or activated partial thromboplastin time < 1.5 × ULN
11. Recovery, to Grade 0-1, from adverse events related to prior anticancer therapy

Exclusion Criteria:

1. Prior therapy with anti PD-L1/TGFβRⅡ targeting treatment.
2. Symptomatic primary central nervous system (CNS) tumor of CNS metastases.
3. Uncontrolled hypertension.
4. Significant thrombotic or hemorrhagic events.
5. Prior CAR-T therapy
6. Severe cardiovascular disease.
7. Active infection requiring therapy
8. Active HIV, hepatitis B or hepatitis C virus
9. Active tuberculosis
10. Anticancer therapy or radiation therapy within 5 half-lives or 4 weeks (whichever is shorter) prior to study entry
11. Pregnant or breast-feeding females
12. Active or history of autoimmune disease or inflammatory disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
To evaluate the incidence and frequency of adverse events following intravenous (IV) infusion of BJ-005 in patients with advanced solid tumor or lymphoma. The assessment will be conducted per CTCAE 5.0 throughout the conduct of the study. | 60 days after the last dose
To determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) of BJ-005 following IV infusion in patients with advanced solid tumor or lymphoma. | 60 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Vicky Gao, MD, Study Director — BJ Bioscience, Inc.
Locations (6):
- United States (6):
  - Mayo Clinic - Phoenix, Phoenix, Arizona
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Hematology/Oncology Assoc. of the Treasure Coast, Port Saint Lucie, Florida
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Carolina BioOncology, Huntersville, North Carolina
  - Next Oncology, Austin, Texas